CLINICAL TRIAL: NCT05479357
Title: Carbetocin Versus Oxytocin for Prophylaxis Against Atonic Primary Post-partum Hemorrhage in High-risk Patients in Sohag University Hospital: A Randomized Controlled Clinical Trial
Brief Title: Carbetocin Versus Oxytocin for Prophylaxis Against Atonic Primary Post-partum Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eman Mahmoud Sabry, Dr., Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Soh-Med-22-07-02
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Atonic Postpartum Hemorrhage; High Risk Pregnancy
Keywords: Atonic Postpartum Hemorrhage; Carbetocin; Oxytocin; High Risk Pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial (Simple randomization)
Who Masked: Participant
Masking Description: Patient will be blinded to the drug to be used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Active Comparator): the control group will be given 10 iu intravenously.
  Interventions: Drug: Oxytocin
- Carbetocin (Active Comparator): the treatment group will be given 100 microgram intravenously.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin — 10 iu will be given intravenously.
  Arms: Oxytocin
Drug: Carbetocin — 100 micrograms will be given intravenously.
  Arms: Carbetocin

SUMMARY:
Comparison between Carbetocin and Oxytocin as prophylaxis against Primary Postpartum Hemorrhage.

DETAILED DESCRIPTION:
Patients will be allocated randomly by simple randomization into either 1- the control group which will be given 10 IU oxytocin intravenously, OR 2- the treatment group which will be given 100 micrograms of carbetocin intravenously.

The trial will be conducted on patients with high risk of developing atonic primary postpartum hemorrhage. The trial will be single blinded. All patients fulfilling the inclusion criteria undergoing elective Caesarean section will be approached by the treating physician and will be asked to participate in the study. An informed written consent will be taken from each patient. The data collected will include base line characteristics such as age, parity, body mass index, the risk for Postpartum hemorrhage in each patient, amount of blood loss, blood units given, complete blood picture (pre and post operative) and coagulation profile.

ELIGIBILITY:
Inclusion Criteria:

* • High risk patients for post-partum hemorrhage who will subjected to Caeserean section either elective or in labour at or after 36 weeks of gestation. This should include one or more of the following:

  1. History of postpartum hemorrhage.
  2. Delivery of a macrosomic baby (> 4000 g).
  3. Multiple gestation.
  4. Polyhydramnios.
  5. Grand Multiparity.
  6. Interstitial or submucous fibroid. (Single larger than 4 cm or Multiple myomata)
  7. Chorioamnionitis.

Exclusion Criteria:

* • Patients without high risk for post-partum hemorrhage.

  * Patients at high risk for postpartum hemorrhage but will deliver vaginally.
  * Patients with medical disorders complicating pregnancy.
  * Patients with coagulation defects.
  * Preterm pregnancies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-28 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Amount of Postpartum Hemorrhage | First 24 hours after Delivery
  Amount of Blood Loss in milliliters. Pre-operative patient's Hemoglobin (Hb) level and 24 hours post-operative will be assessed to quantify amount of blood loss. Additionally, all towels prepared for CS will weighed, and the weight will be marked on each pack before autoclaving. All towels (used and unused) will be weighed again after use, and a difference of 1 gm will be considered as equivalent to 1 mL of absorbed blood.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy M Ameen, MD, Principal Investigator — Faculty of Medicine, Sohag University; Ahmed T Ahmed, MD, Principal Investigator — Faculty of Medicine, Sohag University; Amr O Abdelkareem, MD, Principal Investigator — Faculty of Medicine, Sohag University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waterstone M, Bewley S, Wolfe C. Incidence and predictors of severe obstetric morbidity: case-control study. BMJ. 2001 May 5;322(7294):1089-93; discussion 1093-4. doi: 10.1136/bmj.322.7294.1089. PMID 11337436
- [Background] Zhang WH, Alexander S, Bouvier-Colle MH, Macfarlane A; MOMS-B Group. Incidence of severe pre-eclampsia, postpartum haemorrhage and sepsis as a surrogate marker for severe maternal morbidity in a European population-based study: the MOMS-B survey. BJOG. 2005 Jan;112(1):89-96. doi: 10.1111/j.1471-0528.2004.00303.x. PMID 15663404
- [Background] Dahlke JD, Mendez-Figueroa H, Maggio L, Hauspurg AK, Sperling JD, Chauhan SP, Rouse DJ. Prevention and management of postpartum hemorrhage: a comparison of 4 national guidelines. Am J Obstet Gynecol. 2015 Jul;213(1):76.e1-76.e10. doi: 10.1016/j.ajog.2015.02.023. Epub 2015 Feb 28. PMID 25731692
- [Background] Mantel GD, Buchmann E, Rees H, Pattinson RC. Severe acute maternal morbidity: a pilot study of a definition for a near-miss. Br J Obstet Gynaecol. 1998 Sep;105(9):985-90. doi: 10.1111/j.1471-0528.1998.tb10262.x. PMID 9763050
- [Background] Brace V, Penney G, Hall M. Quantifying severe maternal morbidity: a Scottish population study. BJOG. 2004 May;111(5):481-4. doi: 10.1111/j.1471-0528.2004.00101.x. PMID 15104614
- [Background] Nyflot LT, Sandven I, Stray-Pedersen B, Pettersen S, Al-Zirqi I, Rosenberg M, Jacobsen AF, Vangen S. Risk factors for severe postpartum hemorrhage: a case-control study. BMC Pregnancy Childbirth. 2017 Jan 10;17(1):17. doi: 10.1186/s12884-016-1217-0. PMID 28068990
- [Background] Girault A, Deneux-Tharaux C, Sentilhes L, Maillard F, Goffinet F. Undiagnosed abnormal postpartum blood loss: Incidence and risk factors. PLoS One. 2018 Jan 10;13(1):e0190845. doi: 10.1371/journal.pone.0190845. eCollection 2018. PMID 29320553
- [Background] Nyflot LT, Stray-Pedersen B, Forsen L, Vangen S. Duration of labor and the risk of severe postpartum hemorrhage: A case-control study. PLoS One. 2017 Apr 6;12(4):e0175306. doi: 10.1371/journal.pone.0175306. eCollection 2017. PMID 28384337
- [Background] Maher MA, Sayyed TM, Elkhouly NI. Different routes and forms of uterotonics for treatment of retained placenta: a randomized clinical trial. J Matern Fetal Neonatal Med. 2017 Sep;30(18):2179-2184. doi: 10.1080/14767058.2016.1242124. Epub 2016 Oct 19. PMID 27677547
- [Background] Lawrie TA, Rogozinska E, Sobiesuo P, Vogel JP, Ternent L, Oladapo OT. A systematic review of the cost-effectiveness of uterotonic agents for the prevention of postpartum hemorrhage. Int J Gynaecol Obstet. 2019 Jul;146(1):56-64. doi: 10.1002/ijgo.12836. Epub 2019 May 20. PMID 31049950
- [Background] Withanathantrige M, Goonewardene M, Dandeniya R, Gunatilake P, Gamage S. Comparison of four methods of blood loss estimation after cesarean delivery. Int J Gynaecol Obstet. 2016 Oct;135(1):51-5. doi: 10.1016/j.ijgo.2016.03.036. Epub 2016 Jul 4. PMID 27451396
- [Background] Chong YS, Su LL, Arulkumaran S. Current strategies for the prevention of postpartum haemorrhage in the third stage of labour. Curr Opin Obstet Gynecol. 2004 Apr;16(2):143-50. doi: 10.1097/00001703-200404000-00008. PMID 15017343